CLINICAL TRIAL: NCT03809390
Title: Effects of Vaginal Seeding on Infants' Body Mass Index and Allergy Risk for Caesarean-delivered Children: A Randomized Controlled Study
Brief Title: Effects of Vaginal Seeding on Infants' Body Mass Index and Allergy Risk for Caesarean-delivered Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Liuyang Maternal and Child Health Care Hospital (Unknown)
Responsible Party: Principal Investigator, Jianmeng Liu, Professor in Perinatal Epidemiology, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NSFC.81701538
Record Dates: First submitted 2018-11-17; First posted 2019-01-18 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Overweight and Obesity; Allergy
Keywords: Body mass index; Allergic risk; Vaginal seeding; Randomized controlled study; Caesarean delivery; Overweight and obesity
MeSH Terms: conditions — Overweight; Obesity; Hypersensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal seeding group (Experimental): Swabbing infants born by C-section with a gauze incubated in the maternal vagina about an hour before the C-section. The gauze will be extracted prior to the C-section, kept in a sterile container in an incubator (37 ℃), and taken out from the incubator immediately before the swabbing. The infant will be swabbed with the gauze, starting from the lips, followed by the face, thorax, arms, legs, genitals and anal region, and finally the back. The swabbing will take around 15-20 seconds.
  Interventions: Procedure: Vaginal seeding
- Control group (No Intervention): Managed based on the standard practice in the study site

INTERVENTIONS:
Procedure: Vaginal seeding — The same as that stated in arm descriptions.
  Arms: Vaginal seeding group

SUMMARY:
This is a single-blind randomized controlled trial, aiming to evaluate the effects of vaginal seeding on body mass index as well as allergy risk for cesarean-delivered infants. It will be conducted in Liuyang city of China, and the targeted sample size is 106. All the eligible pregnant women will be randomly assigned to either the intervention or control group, and their babies of the participants will be followed up to 24 months of age.

DETAILED DESCRIPTION:
Many studies have suggested that caesarean-delivered children are at higher risks of developing metabolic and allergic diseases like obesity and asthma, possibly because newborns born by caesarean section were lack of exposure to maternal vaginal flora. It is needed to explore a simple, convenient, and safe intervention strategy to reduce caesarean-related risks. In a recent non-randomized study, the authors found that exposure of caesarean-delivered newborns to maternal vaginal fluid at birth (i.e., vaginal seeding) could partially restore the microbiota of them at 30 days after births, but the long-term health consequences of restoring the microbiota of caesarean-delivered infants remain unclear.

In this randomized study, the investigators aim to examine whether the changes in newborns' microbiota will persist to 24 month of age, and whether vaginal seeding will have any effects on body mass index and allergy risk from birth to 24 months of age. the investigators will enroll a total of 106 pregnant women, and the participants' infants will be followed up at 0 (before hospital discharge), 6, 12, 18 and 24 months. At each follow-up visit, a questionnaire survey including information on feeding, medication, and allergic status will be conducted, infants' height and weight will be measured, and feces will be collected. At 18-month-old visit, infants' venous blood will be also collected for the assay of multiallergen. The primary outcomes were body mass index and allergy risk index. The secondary outcomes included the microbiota profile, allergic symptoms and diseases, overweight/obesity, and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* local resident in Liuyang city
* Singleton, term pregnancy (≥37 weeks of gestation)
* Cesarean section before labor starts without maternal complications, or cesarean section after the start of labor but the cervix is less than 3 cm
* Vaginal pH< 4.5 at enrollment

Exclusion Criteria:

* Positive testing for HIV, HBV, syphilis or GBS infection at gestation
* Vaginal infections such as genital herpetic lesions or chlamydia
* Bacterial vaginosis
* Trichomonas or fungous in leucorrhea
* Pregnant women or her spouse with severe allergic diseases, such as asthma and severe drug allergy
* Vaginal pH ≥4.5 at 1-2 hours before the cesarean section
* Other conditions not suitable for intervention as judged by obstetricians

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2018-11-17 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
infant's body mass index | At 6 months
  Body mass index in original scale and z-score
infant's body mass index | At 12 months
  Body mass index in original scale and z-score
infant's body mass index | At 18 months
  Body mass index in original scale and z-score
infant's body mass index | At 24 months
  Body mass index in original scale and z-score
infant's allergy risk score | At 18 months after birth
  Calculated based on the measurements of multiallergens with 0-6 classes,higher values represent a worse outcome which means more susceptible to allergic diseases

SECONDARY OUTCOMES:
Infants' gut microbiota profile | At baseline (Meconium), 6, 12 ,18 and 24 months after birth
  Intestinal flora will be detected by 16sRNA sequencing using feces samples
Rate of overweight/obesity | At 6, 12 ,18 and 24months
  Defined by body mass index
Rate of allergic symptoms and common allergic diseases | At 61, 12 ,18 and 24 months
  Collected by using a structured questionnaire
Rate of adverse effects | From birth to 24 months
  Infection-related diseases and others

CONTACTS AND LOCATIONS:
Overall Officials: Jian-meng Liu, PhD, Study Chair — Peking University; Hong-tian Li, PhD, Principal Investigator — Peking University; Shujin Zhou, MD, Study Director — Liuyang Maternal and Child Health Care Hospital; Yang Liu, PhD Candidate, Study Director — Peking University
Locations (1):
- Liuyang Maternal and Child Health Care Hospital, Guankou, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared upon the request of other researchers, and all the key variables that will be reported in the main paper are planned to be shared
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: After the publication of the main paper (hopefully before the end of 2022), the data will be available to share to other researchers
Access Criteria: Researchers should request the data via the following Email: lihongtian@pku.edu.cn or liujm@pku.edu.cn